CLINICAL TRIAL: NCT00005737
Title: Tuberculosis Prophylaxis in the Homeless--A Controlled Trial
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4946; R01HL055729 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-04

CONDITIONS: Lung Diseases; Tuberculosis
MeSH Terms: conditions — Lung Diseases; Tuberculosis

SUMMARY:
To conduct a three-arm, randomized controlled trial of methods to improve adherence to biweekly directly observed prophylaxis (DOPT) for tuberculosis in homeless adults in San Francisco.

DETAILED DESCRIPTION:
BACKGROUND:

Tuberculosis was on the decline from the mid 1950s until the mid 1980s; however, the United States is now experiencing a resurgence of tuberculosis. In 1992, approximately 27,000 new cases were reported, an increase of about 20 percent from 1985 to 1992. Not only are tuberculosis cases on the increase, but a serious aspect of the problem is the recent occurence of outbreaks of multidrug resistant (MDR) tuberculosis, which poses an urgent public health problem and requires rapid intervention.

Control programs involve two major components. First, and of highest priority, is to detect persons with active tuberculosis and treat them with effective antituberculosis drugs, which prevents death from tuberculosis and stops the transmission of infection to other persons. Treatment of active tuberculosis involves taking multiple antituberculosis drugs daily or several times weekly for at least six months. Failure to take the medications for the full treatment period may mean that the disease is not cured and may recur. If sufficient medications are not prescribed early and taken regularly, the tuberculosis organism can become resistant to the drugs, and the drug resistant tuberculosis then may be transmitted to other persons. Drug resistant disease is difficult and expensive to treat, and in some cases, cannot be treated with available medications.

The second major goal of control efforts is the detection and treatment of persons who do not have active tuberculosis, but who have latent tuberculosis infection. These people may be at high risk of developing active tuberculosis. The only approved treatment modality for preventive therapy requires treatment daily or twice weekly for a minimum of six months, and many patients do not complete the full course of therapy. Public and patient programs are needed to increase the awareness of the problems associated with tuberculosis control.

The study is part of the NHLBI initiative "Behavioral Interventions for Control of Tuberculosis" . The concept for the initiative originated from the National Institutes of Health Working Group on Health and Behavior. The Request for Applications was released in October, 1994.

DESIGN NARRATIVE:

Three approaches were compared for improving adherence to biweekly directly observed prophylaxis for tuberculosis in the homeless: $5 biweekly money incentive (MI) for adherence to DOPT, $5 value biweekly non-money incentive (NMI) for adherence to DOPT, and $5 biweekly money incentive supplemented by a peer community outreach worker (MI + PCOW). The outreach worker assisted subjects with completion of adherence to DOPT. Predictors of adherence to DOPT were examined, including sociodemographic, psychological and behavioral, and environmental factors.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 1999-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Moss — University of California

REFERENCES:
- [Background] Bangsberg D, Tulsky JP, Hecht FM, Moss AR. Protease inhibitors in the homeless. JAMA. 1997 Jul 2;278(1):63-5. No abstract available. PMID 9207341
- [Background] Tulsky JP, Hahn JA, Long HL, Chambers DB, Robertson MJ, Chesney MA, Moss AR. Can the poor adhere? Incentives for adherence to TB prevention in homeless adults. Int J Tuberc Lung Dis. 2004 Jan;8(1):83-91. PMID 14974750